CLINICAL TRIAL: NCT06033495
Title: Myocardial Ischemia by 15O-H2O PET/CT in Patients With Coronary Artery Disease and Refractory Angina - Evaluation of the Coronary Sinus Reduction Stent Method
Brief Title: Myocardial Ischemia After Coronary Sinus Reduction Stent Implantation
Acronym: MICS-Reduce
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Øyvind Lie, Principal Investigator, Oslo University Hospital
Other Study IDs: 657796
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with refractory angina undergoing coronary sinus reduction stent implantation
  Interventions: Device: Coronary sinus reduction stent

INTERVENTIONS:
Device: Coronary sinus reduction stent — Percutaneous stent implantation to reduce the dimension of the coronary sinus

SUMMARY:
Chronic angina pectoris refractory to medical and revascularization therapies is a disabling medical condition and a major public health problem. Patients with refractory angina have limited treatment options. One proposed therapy modality is transcatheter implantation of a reduction stent in the coronary sinus. Coronary sinus reduction stents have been shown to reduce angina burden considerably and to improve quality of life. The reduction stent is assumed to increase myocardial perfusion and reduce myocardial ischemia, but the mechanism of action is poorly understood.

The aim of this project is to assess the myocardial ischemia burden in patients with refractory angina who are undergoing a transcatheter coronary sinus reducer procedure. This is a clinical non-randomized self-controlled cohort study with blinded outcome adjudication for changes in myocardial perfusion. Patients with refractory angina will be systematically examined before implantation of the coronary sinus reduction stent and after 6 months. The primary outcome, changes in myocardial perfusion on the gold standard 15O-H2O PET/CT will be evaluated on blinded perfusion scans where the stent is invisible. To provide context to the findings, we will also evaluate whether changes in myocardial ischemia are associated with less angina and better cardiac function parameters. Effects of stent implantation on angina symptoms and quality of life could be affected by a placebo effect.

Treatment options for patients with refractory angina is needed, and results from the present study will explore if coronary sinus reduction stents are improving myocardial ischemia in this patient group. Signs of improved objective perfusion will inspire confidence in the method.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease and refractory angina
* Clinical indication for coronary sinus reduction stent implantation
* Written informed consent
* Anticipated compliance with protocol

Exclusion Criteria:

* Ineligibility for coronary sinus reduction stent implantation
* Lack of informed consent
* Not expected to comply with protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease and refractory angina who are under clinical care are informed and screened for participation if consent is provided.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial ischemia | 6 months
  Change in myocardial flow reserve on 15O-H2O PET/CT

SECONDARY OUTCOMES:
Change in angina burden | 6 months
  Seattle angina questionnaire (SAQ-7) score ranging 0 (bad) -100 (good) will be assessed at baseline and after 6 months.
Change in quality of life | 6 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) score ranging 0 (bad) -100 (good) will be assessed at baseline and after 6 months.
Change in exercise capacity | 6 months
  Maximum oxygen extraction on cardiopulmonary exercise test assessed at baseline and after 6 months.
Change in coronary microcirculation | 6 months
  Invasive assessment of coronary flow reserve (CFR) at baseline and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind H Lie, Principal Investigator — Oslo University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
We aim to share data upon request from other academic investigators, but await EC approval